CLINICAL TRIAL: NCT03956953
Title: A Randomized, Double-Blind, Placebo-Controlled, Single- And Multiple-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BMS-986165 in Healthy Chinese Subjects
Brief Title: Single and Multiple Dose Pharmacokinetics of BMS-986165 in a Randomized, Double-Blind, Placebo-Controlled Study in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM011-053
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases | interventions — deucravacitinib

STUDY DESIGN:
Intervention Model Description: There will be two dose groups. Once the safety and tolerability up to discharge (Day 24) of Group 1, has been assessed and deemed safe; dosing for Group 2 will begin.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group 1: BMS-986165 Dose 1 (Experimental): Participants will receive Dose 1 on Day 1, and from Day 5 - 19.
  Interventions: Drug: BMS-986165
- Group 2: BMS-986165 Dose 2 (Experimental): Participants will receive Dose 2 on Day 1, and from Day 5 - 19.
  Interventions: Drug: BMS-986165
- Group 1: Placebo Dose 1 (Placebo Comparator): Participants will receive placebo matching Dose 1 on Day 1, and from Day 5 - 19.
  Interventions: Other: Placebo
- Group 2: Placebo Dose 2 (Placebo Comparator): Participants will receive placebo matching Dose 2 on Day 1, and from Day 5 - 19.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986165 — Dose 1 or Dose 2 on Day 1, and from Days 5-19'
  Arms: Group 1: BMS-986165 Dose 1; Group 2: BMS-986165 Dose 2
Other: Placebo — Placebo matching Dose 1 or Dose 2 on Day 1, and from Days 5-19
  Arms: Group 1: Placebo Dose 1; Group 2: Placebo Dose 2

SUMMARY:
Main objective of this study is to assess BMS-986165 plasma PK following single and multiple oral doses of BMS-986165 in healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent.
* Healthy participants, as determined by physical examination, ECGs, and clinical laboratory and procedure determinations.
* Body mass index (BMI) of 18 to 24 kg/m2, inclusive, and total body weight >= 50 kg.

Exclusion Criteria:

* History of allergy to drug class or related compounds.
* History or evidence of active infection within 7 days of study day 1.
* Drug or alcohol abuse within 6 months of study treatment administration.

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of BMS-986165 | Days 1 to 4, Day 5, and Day 19
Time to Maximum Observed Plasma Concentration (Tmax) of BMS-986165 | Days 1 to 4, Day 5, and Day 19
Area Under The Plasma Concentration-Time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC(0-T)) of BMS-986165 | Days 1 to 4, Day 5, and Day 19
Area Under The Plasma Concentration-Time Curve From Time Zero Extrapolated To Infinite Time (AUC(INF)) of BMS-986165 | Day 1 to Day 4
Apparent Plasma Elimination Half-Life (T-HALF) of BMS-986165 | Days 1 to 4, Day 5, and Day 19
Apparent Oral Total Body Clearance (CLT/F) of BMS-986165 | Days 1 to 4, Day 5, and Day 19
Metabolic Ratio for AUC(INF) of Metabolite (BMT-153261 and BMT-158170) Over Parent (BMS-986165) - MR(AUC[INF]) | Day 1 to Day 4
Metabolic Ratio for Cmax of Metabolite (BMT-153261 and BMT-158170) Over Parent (BMS-986165) - MR(Cmax) | Days 1 to 4, Day 5, and Day 19
Apparent Volume of Distribution (Vz/F) of BMS-986165 | Days 1 to 4, Day 5, and Day 19
Time to Maximum Observed Plasma Concentration (Tmax) of BMS-986165 | Day 5 to Day 19
Area Under the Plasma Concentration-Time Curve in a Dosing Interval (AUC(TAU)) of BMS-986165 | Day 5 and Day 19
Effective Elimination Half-Life (T-HALFeff) of BMS-986165 | Days 1 to 4, Day 5, and Day 19
Trough Observed Plasma Concentration (Ctrough) of BMS-986165 | Day 2 to 20
Average Plasma Concentration at Steady State (Css-avg) of BMS-986165 | Days 1 to 4, Day 5, and Day 19
Accumulation Index (AI) of BMS-986165 | Days 1 to 4, Day 5, and Day 19
Metabolic Ratio for AUC(TAU) of Metabolite (BMT-153261 and BMT-158170) Over Parent (BMS-986165) - MR(AUC[TAU]) | Day 5 to Day 19
Degree of Fluctuation (DF) of BMS-986165 | Days 1 to 4, Day 5, and Day 19

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to Day 31
Number of Participants With Clinically Significant Change in Clinical Laboratory Values | Up to Day 24
Number of Participants With Clinically Significant Change in Vital Signs | Up to Day 24
Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) | Up to Day 24
Number of Participants With Clinically Significant Change in Physical Examination | Up to Day 24
Maximum Observed Plasma Concentration (Cmax) of Metabolites BMT-153261 and BMT-158170 | Days 1 to 4, Day 5, and Day 19
Time to Maximum Observed Plasma Concentration (Tmax) of B Metabolites BMT-153261 and BMT-158170 | Days 1 to 4, Day 5, and Day 19
Area Under The Plasma Concentration-Time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC(0-T)) of Metabolites BMT-153261 and BMT-158170 | Days 1 to 4, Day 5, and Day 19
Area Under The Plasma Concentration-Time Curve From Time Zero Extrapolated To Infinite Time (AUC(INF)) of Metabolites BMT-153261 and BMT-158170 | Days 1 to 4, Day 5, and Day 19
Apparent Plasma Elimination Half-Life (T-HALF) of Metabolites BMT-153261 and BMT-158170 | Days 1 to 4, Day 5, and Day 19
Area Under the Plasma Concentration-Time Curve in a Dosing Interval (AUC(TAU)) of Metabolites BMT-153261 and BMT-158170 | Days 1 to 4, Day 5, and Day 19
Effective Elimination Half-Life (T-HALFeff) of Metabolites BMT-153261 and BMT-158170 | Days 1 to 4, Day 5, and Day 19
Trough Observed Plasma Concentration (Ctrough) of Metabolites BMT-153261 and BMT-158170 | Days 1 to 4, Day 5, and Day 19
Average Plasma Concentration at Steady State (Css-avg) of Metabolites BMT-153261 and BMT-158170 | Days 1 to 4, Day 5, and Day 19
Accumulation Index (AI) of Metabolites BMT-153261 and BMT-158170 | Days 1 to 4, Day 5, and Day 19
Degree of Fluctuation (DF) of Metabolites BMT-153261 and BMT-158170 | Days 1 to 4, Day 5, and Day 19
Total Amount of Drug Recovered in Urine (URt) Following Single Oral Doses of BMS-986165 | Day 1 to Day 5
Total Percent of Administered Dose Recovered Unchanged in Urine (%URt) Following Single Oral Doses of BMS-986165 | Day 1 to Day 5
Renal Clearance (CLR) Following Single Oral Doses of BMS-986165 | Day 1 to Day 5

CONTACTS AND LOCATIONS:
Locations (1):
- Local Institution, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Jing S, Lin Y, Dockens R, Marchisin D, He B, Girgis IG, Chimalakonda A, Murthy B, Aras U. Pharmacokinetics and Safety of the Tyrosine Kinase 2 Inhibitor Deucravacitinib in Healthy Chinese Subjects. Dermatol Ther (Heidelb). 2023 Dec;13(12):3153-3164. doi: 10.1007/s13555-023-01050-7. Epub 2023 Nov 19. PMID 37981596
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm